CLINICAL TRIAL: NCT00079053
Title: A Phase I Study of Adjuvant OSI-774 (Tarceva®) in Patients Following Combined Chemo-Radiotherapy for Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Brief Title: Adjuvant Erlotinib After Completing Chemoradiotherapy in Locally Advanced Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN5; CAN-NCIC-HN5 (Other: PDQ); ROCHE-CAN-NCIC-HN5 (Other: Roche); CDR0000353485 (Other: PDQ)
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; salivary gland squamous cell carcinoma; stage III salivary gland cancer; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — Erlotinib Hydrochloride; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: erlotinib hydrochloride
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Giving erlotinib after chemoradiotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of adjuvant erlotinib when given after completing chemoradiotherapy in treating patients with locally advanced squamous cell carcinoma (cancer) of the head and neck.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the recommended dose of adjuvant erlotinib after the completion of chemoradiotherapy in patients with stage III, IVA, or IVB squamous cell carcinoma of the head and neck.
* Determine the toxicity of this drug in these patients.
* Determine the effects of this drug on plasma and urinary angiogenic factors (specifically vascular endothelial growth factor receptor [VEGFR], VEGFR1, VEGFR2, and basic fibroblast growth factor levels) in these patients.
* Compare the disease-free survival of patients treated with this drug after chemoradiotherapy vs historical control patients treated with chemoradiotherapy alone.
* Correlate levels of angiogenic factors with initial blood vessel concentration in the tumor and the presence or absence of EGFRvIII mutation in patients treated with this drug.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive oral erlotinib once daily on days 1-28. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 6 patients receive escalating doses of erlotinib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, an additional 8 patients are treated at that dose level.

Patients are followed at 4 weeks, every 12 weeks for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 6-20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed squamous cell carcinoma of the head and neck

  * Stage III, IVA, or IVB
* Must have completed cisplatin- or carboplatin-based chemoradiotherapy within the past 4-12 weeks

  * Prior radiotherapy must have been given with a radical intent with receipt of at least 90% of planned dose
* No evidence of disease or presence of inoperable minimal residual disease, defined by 1 of the following:

  * Complete response at primary tumor site and nodes (with or without nodal surgery after chemoradiotherapy)
  * Negative lymph node status (by physical or radiological exam) AND persistent tumefaction less than 25% of original tumor size or residual mass due to scarring
* Tumor tissue samples available for EGFRvIII mutation analysis
* No known brain metastasis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* ALT/AST < 2 times upper limit of normal (ULN)
* Bilirubin < ULN (unless due to Gilbert's syndrome)

Renal

* Creatinine < 1.5 times ULN

Cardiovascular

* No myocardial infarction within the past year
* No cardiac ventricular arrhythmias requiring medication
* No history of cardiac disease
* No uncontrolled high blood pressure
* No unstable angina
* No congestive heart failure

Ophthalmic

* No history of severe dry eye syndrome, Sjögren's syndrome, or keratoconjunctivitis sicca
* No severe exposure keratopathy
* No abnormal slit-lamp examination using a vital dye (e.g., fluorescein or Bengal-Rose)
* No abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* No disorder that might increase the risk for epithelium-related complication (e.g., bullous keratopathy, aniridia, severe chemical burns, or neutrophilic keratitis)
* No congenital abnormality (e.g., Fuch's dystrophy)
* No ocular inflammation or infection

Gastrointestinal

* Able to take oral medication
* No gastrointestinal (GI) tract disease requiring IV alimentation
* No uncontrolled inflammatory GI disease (e.g., Crohn's disease or ulcerative colitis)
* No active peptic ulcer disease

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious active infection
* No other serious underlying medical condition that would preclude study participation
* No prior allergic reaction to compounds of similar chemical or biological composition to erlotinib
* No other malignancy with the past 5 years except adequately treated non-melanoma skin cancer (unless in the same area treated with radical radiotherapy) or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* Recovered from prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* Recovered from prior radiotherapy

Surgery

* See Disease Characteristics
* No prior surgical procedure affecting absorption
* No concurrent ophthalmic surgery

Other

* More than 4 weeks since other prior investigational drugs
* No other concurrent investigational agents
* No other concurrent anticancer therapy
* Concurrent oral anticoagulants (e.g., warfarin) allowed provided there is increased vigilance with respect to INR
* Concurrent nasogastric or gastrostomy tube feeding for dysphagia allowed provided there is no evidence of significant residual mucositis (i.e., > grade 1)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-03-02 (Actual); Primary Completion 2008-12-09 (Actual); Study Completion 2011-01-18 (Actual)

PRIMARY OUTCOMES:
Toxicity/feasibility assessed by NCI CTC v2.0 at the end of course 1
Recommended phase II dose at the end of course 1

SECONDARY OUTCOMES:
Correlative studies (archival and prospective) at accrual completion
Disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Denis Soulieres, MD, MSC, Study Chair — CHUM - Hotel Dieu Hospital
Locations (2):
- Canada (2):
  - London Regional Cancer Program, London
  - CHUM - Hopital Notre-Dame, Montreal

IPD SHARING:
Plan to Share IPD: No